CLINICAL TRIAL: NCT05211232
Title: A Phase III, Double-Blind, Placebo-Controlled Study of Neoadjuvant Tislelizumab + Chemotherapy Followed by Adjuvant Tislelizumab for the Treatment of Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Neoadjuvant and Adjuvant Tislelizumab for Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Hospital of Guizhou Province (Other); Hunan Cancer Hospital (Other); Wuzhou Red Cross Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-FXY-452
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP combined with Tislelizumab neoadjuvant therapy+CCRT+Tislelizumab adjuvant therapy (Experimental): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on day 1,8) , cisplatin (80mg per square meter on day 1) and tislelizumab(200mg) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1,D22,D43 of RT) ,then followed by adjuvant therapy with tislelizumab(200mg) every three weeks for eight cycles after radiotherapy
  Interventions: Drug: Tislelizumab
- GP combine with Placebo neoadjuvant therapy+CCRT+Placebo adjuvant therapy (Placebo Comparator): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on day 1,8) , cisplatin (80mg per square meter on day 1) and Placebo(200mg) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1,D22,D43 of RT) ,then followed by adjuvant therapy with Placebo(200mg) every three weeks for eight cycles after radiotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tislelizumab — GP combine with Tislelizumab neoadjuvant therapy+CCRT+Tislelizumab adjuvant therapy
  Other Names: BGB-A317
  Arms: GP combined with Tislelizumab neoadjuvant therapy+CCRT+Tislelizumab adjuvant therapy
Drug: Placebo — GP combine with Placebo neoadjuvant therapy+CCRT+Tislelizumab adjuvant therapy
  Arms: GP combine with Placebo neoadjuvant therapy+CCRT+Placebo adjuvant therapy

SUMMARY:
The purpose of this study is to explore the efficacy and safety of a combination of GP chemotherapy and tislelizumab in neoadjuvant therapy combined with tislelizumab in adjuvant therapy of locoregionally advanced nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Platinum-based concurrent chemoradiotherapy is the standard of care for patients with locoregionally advanced nasopharyngeal carcinoma(NPC). Gemcitabine plus cisplatin(GP) has been demonstrated an effective chemotherapy regimen for NPC patients in previous studies. The results of GP combined with concurrent chemoradiotherapy in the treatment of locoregionally advanced nasopharyngeal carcinoma showed 10% of locoregionally advanced NPC patients had complete response after three cycles of GP neoadjuvant chemotherapy, and GP neoadjuvant chemotherapy added to chemoradiotherapy significantly improved recurrence-free survival (85.3% vs 76.5%) and overall survival (94.6% vs 90.3%) among locoregionally advanced NPC patients , as compared with chemoradiotherapy alone. Therefore, GP regimen has been established as the highest level of evidence-based neoadjuvant chemotherapy in the 2020 National Comprehensive Cancer Network (NCCN) guidelines. Recently, immune checkpoint inhibitors, such as anti-programmed cell death-1 (PD-1)monoclonal antibody has shown promising efficacy in the treatment of tumor patients. Clinical trials have shown objective response rates of 20.5%-34% in patients with recurrent or metastatic NPC patients receiving anti PD-1 monoclonal antibody immunotherapy including pembrolizumab, nivolumab, camrelizumab, and toripalimab. The current NCCN guidelines recommend anti PD-1 monoclonal antibody as a second-line treatment for recurrent or metastatic NPC. More and more evidence show that immunotherapy combined with chemotherapy has a synergistic effect in treating tumors. GP chemotherapy combined with anti PD-1 antibody has achieved the initial effect in NPC. Phase 1 trials have shown the combination of camrelizumab plus GP chemotherapy in recurrent or metastatic NPC led to a proportion of 91% patients achieving an objective response. In addition, previous studeis showed that PD-1 antibody adjuvant therapy had good feasibility and effectiveness in the treatment of nasopharyngeal carcinoma. Tislelizumab, approved by the National Medical Products Administration in China, is an anti-PD-1 monoclonal IgG4 antibody with higher affinity to PD-1 than pembrolizumab and nivolumab and was engineered to minimize binding to FcγR on macrophages in order to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. Multiple clinical trials have shown strong anti-neoplastic activity of tislelizumab in various tumors including NPC. Clinical trial has shown an objective response rates of 43% in patients with recurrent metastatic nasopharyngeal carcinoma treated with tirelizumab, which is superior to other anti PD-1 monoclonal antibodys. So we hypothesize that GP neoadjuvant chemotherapy combined with tislelizumab and tislelizumab adjuvant therapy could further improve survival of patients with locaregionally advanced NPC. Based on this, this study aims to evaluate the efficacy and safety of gemcitabine plus cisplatin chemotherapy combined with tislelizumab neoadjuvant therapy, followed by cisplatin based concurrent chemoradiotherapy, then followed by tislelizumab adjuvant therapy in the patients with locoregionally advanced nasopharyngeal carcinoma, to provide new evidence for individualized comprehensive treatment in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent.
2. Age ≥ 18 years and ≤70 years,men or non-pregnant women.
3. Patients with histologically confirmed Nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type, WHO II or III).
4. Tumor staged as III-IVA (AJCC 8th, except T3N0，T3N1(Only retropharyngeal lymph nodes metastasized).
5. No previous anti-tumor treatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
7. Adequate marrow function:White blood cell count (WBC)≥4.0×109 /L, Hemoglobin ≥ 90g/L, Platelet count ≥100×109/L.
8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2×upper limit of normal (ULN),serum total bilirubin (TBIL) ≤2.0 times the upper limit of normal (ULN) .Adequate renal function: creatinine clearance rate≥60 ml/min or Creatinine ≤1.5× upper limit of normal value.

Exclusion Criteria:

1. Patients with recurrent or metastatic nasopharyngeal carcinoma.
2. Histologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
3. Prior therapy with radiation or systemic chemotherapy.
4. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
5. Seropositivity for human immunodeficiency virus (HIV).
6. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Prior exposure to immune checkpoint inhibitors,including anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies.
8. Patients with immunodeficiency disease or a history of organ transplantation.
9. Received large doses of glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressants within 4 weeks.
10. Patients with severe dysfunction of heart, liver, lung, kidney or marrow.
11. Patients with severe, uncontrolled disease or infections.
12. Received other research drugs or in other clinical trials at the same time.
13. Refuse or fail to sign the informed consent .
14. Patients with other treatment contraindications.
15. Patients with personality or mental disorders, incapacity or limited capacity for civil conduct.
16. Hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV deoxyribonucleic acid (HBV DNA) ≥1000cps/ml.
17. Patients with positive HCV antibody test will only be enrolled in this study if the PCR test for HCV RNA is negative.
18. Patients who were known to be intolerable or allergic to treatment drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 9 weeks
  CR assessed by investigator, according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the neoadjuvant therapy. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) .
Progression-free Survival (PFS) | 3 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival(OS) | 3 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
Locoregional failure-free survival(LRRFS) | 3 years
  defined as the time from random assignment to local or regional relapse, or death from any cause.
Distant metastasis-free survival(DMFS) | 3 years
  defined as the time from random assignment to distant metastasis, or death from any cause.
Number of participants with adverse events | up to 3 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: haiqiang Mai, MD, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - The Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Result] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578
- [Result] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638
- [Result] Xu J, Bai Y, Xu N, Li E, Wang B, Wang J, Li X, Wang X, Yuan X. Tislelizumab Plus Chemotherapy as First-line Treatment for Advanced Esophageal Squamous Cell Carcinoma and Gastric/Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2020 Sep 1;26(17):4542-4550. doi: 10.1158/1078-0432.CCR-19-3561. Epub 2020 Jun 19. PMID 32561664